CLINICAL TRIAL: NCT01501344
Title: A 12-week, Open-label Study to Evaluate the Effect of MBP-80 (200g of Yogurt With Fortified Calcium Content and MBP 80 mg) on Bone Remodelling as Assessed by Bone Turnover Markers in Early Postmenopausal Women
Brief Title: Open-label Study to Evaluate the Effect of MBP-80 on Bone Remodelling
Acronym: YogA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe De Recherche En Rhumatologie Et Maladies Osseuses Inc. (Industry)
Collaborators: Aliments ULTIMA Foods Inc. (Industry)
Responsible Party: Principal Investigator, Jacques Brown, Director, Groupe De Recherche En Rhumatologie Et Maladies Osseuses Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010YogA80; MBP-80 and Bone Remodelling (Other: GRMO)
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2011-12

CONDITIONS: Postmenopausal Osteoporosis
Keywords: osteoporosis; postmenopausal women; bone remodelling; bone turnover markers
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: 200 g yogurt with fortified calcium content and MBP 80 mg — Intake of one container of vanilla or strawberry yogurt in the morning on a daily basis during 12 weeks.
  Other Names: Yoplait Asana TM

SUMMARY:
This study will determine if daily oral intake of 200g of a marketed yogurt with fortified calcium content and a milk basic protein (MBP)80 mg benefits on bone cells activity in postmenopausal women. The efficacy of the product is measured by examining the variation of biochemical markers of bone turnover. MBP 80 is a particular protein contained in milk; it has been added to the yogurt provided for this study. The effects of MBP 80 on the quality of bone tissue have not yet been proven.

DETAILED DESCRIPTION:
The morbidity and mortality associated with osteoporotic related fractures is devastating in terms of disability to an individual and cost to the global economy. As the world's population ages, this will present a major public health issue since a larger proportion of women remain undiagnosed and untreated even with the availability of therapies and calcium and vitamin D supplements. Consequently, it remains important to evaluate dairy products (milk, cheese, and yogurt) that can be safely provided as a supplement for bone health in addition to the current pharmacological treatments.

The rationale of this study is to assess the beneficial effect of a daily dietary supplement of MBP 80 mg in a yogurt matrix with fortified calcium content on bone remodelling in healthy early postmenopausal women with neither osteoporosis nor estrogens/progestin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Early postmenopausal women, aged 45-60 yrs old inclusive, with 1-5 yrs since last menses; naturally or surgically menopausal as a result of bilateral oophorectomy. Hysterectomized (≤ 5 yrs) women 50-60 yrs old.
* Lumbar Spine (L.S.;L1-L4) BMD > 0.772 g/cm2 (T-score of -2.5 on Hologic) and,
* Femoral Neck BMD > 0.572 g/cm2 (T-score of -2.5 on Hologic) and,
* Total Hip BMD > 0.637 g/cm2 (T-score of -2.5 on Hologic).
* Subjects must sign the Ethic Committee approved Informed Consent Form before any study procedure is initiated.

Exclusion Criteria:

* Any intake of calcium and vitamin D supplements including multivitamins, nutritional or dietary supplements of any kind containing calcium and vit D within 3 months prior to screening visit 1A.
* Daily dietary calcium intake > 600 mg as assessed by the Calcium Intake Calculator (Appendix E).
* Subjects who already suffer from osteoporosis on the basis of a low BMD T-score ≤ - 2.5 at any site or a personal history of fragility fracture after age 40.
* Any past or present use of:
* Bisphosphonate
* PTH or PTH derivatives, eg. teriparatide
* Androgens, anabolic steroids or testosterone
* Tibolone
* Calcitriol
* Strontium ranelate
* Lithium, chronic warfarin or heparin use > 3 months, anticonvulsants (benzodiazepines are allowed), gonadotrophin-releasing hormone agonists, glitazones.
* Administration of any of the following treatments within the last 3 months prior to screening:
* Glucocorticosteroids (> 5 mg prednisone equivalent per day for > 10 days)
* Systemic hormone replacement therapy
* Selective estrogen receptor modulators (SERMs), eg, raloxifene
* Calcitonin
* Any unapproved hormone-like treatment in the opinion of the Principal Investigator (P.I.), i.e. phytoestrogens, isoflavones, etc.
* Antacids, H2 blockers, proton pump inhibitors for > 10 days
* Iron supplements for > 10 days
* Any condition or disease that may, according to the P.I., interfere with the evaluation of L.S. and Hip BMD; including but not limited to: advanced scoliosis or extensive lumbar fusion, less than 2 lumbar vertebrae (L1-L4) evaluable for DXA.
* Hyper or hypothyroidism: patients on stable dose of thyroid treatment with normal TSH will be allowed. Lab values for TSH must be normal or slightly abnormal, though clinically non significant in the opinion of the P.I.
* Current hyper or hypoparathyroidism, in the opinion of the P.I.
* Current hypocalcemia, in the opinion of the P.I.
* Vit D insufficiency (25-OH vitamin D level < 40 nmol/L)
* Significantly impaired renal function hereby defined as an estimated GFR ≤ 60 mL/min/ 1.73 m2 (4-variable MDRD equation).
* Rheumatoid arthritis.
* Paget's disease of bone.
* Any history of cancer within the past 5 years (except for basal cell carcinoma, dermal squamous cell carcinoma with 6 month remission and cervix carcinoma in situ).
* Any bone disease, i.e. osteomalacia or osteogenesis imperfecta.
* Chronic asthma, in the opinion of the P.I.
* Malabsorption syndrome (coeliac disease, inflammatory bowel disease, gastric bypass).
* Height, weight and girth which may preclude accurate DXA measurement; BMI outside ranges between 18.5 and 35 inclusive.
* Variation of more than 2 kg (gain or loss) within 2 months of the Screening.
* Presence of any vertebral fracture on the screening VFA (Vertebral Fracture Assessment) measured by DXA.
* Any previous or ongoing clinically significant illness that, in the opinion of the P.I., could prevent the patient from completing the study.
* Evidence of alcohol or substance abuse within the last 12 months that the P.I. believes would interfere with understanding or completing the study.
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Median percent change in levels of serum β CTX (sCTX), a bone resorption marker. | 12 weeks
  The primary efficacy variable, the median percent change from baseline (Day 0) in levels of serum β-CTX (sCTX) at week 12, will be compared to the corresponding median percent change from day minus 28 (Day - 28) in levels of serum β-CTX (sCTX) at Day 0 for each participant.

SECONDARY OUTCOMES:
Median percent change in levels of P1NP, a bone formation marker. | 12 weeks
  A secondary efficacy variable, the median percent change from baseline (Day 0) in levels of serum P1NP (sP1NP) at week 12, will be compared to the corresponding median percent change from day minus 28 (Day - 28) in levels of serum P1NP(sP1NP) at Day 0 for each participant.
Median percent change in levels of serum β-CTX (sCTX), a bone resorption marker | 4 weeks
  A secondary efficacy variable, the median percent change from baseline (Day 0) in levels of serum β-CTX(sCTX) at week 4, will be compared to the corresponding median percent change from day minus 28 (Day - 28) in levels of serum β-CTX(sCTX) at Day 0 for each participant.
Median percent change in levels of urinary NTX(uNTX), a bone resorption marker. | weeks 4 and 12
  A secondary efficacy variable, the median percent change from baseline (Day 0) in levels of urinary NTX(uNTX) at weeks 4 and 12, will be compared to the corresponding median percent change from day minus 28 (Day - 28) in levels of urinary NTX(uNTX) at Day 0 for each participant.
Median percent change in levels of serum osteocalcin (sOC), a bone formation marker. | 12 weeks
  A secondary efficacy variable, the median percent change from baseline (Day 0) in levels of serum osteocalcin(sOC) at week 12, will be compared to the corresponding median percent change from day minus 28 (Day - 28) in levels of serum osteocalcin(sOC) at Day 0 for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques P Brown, M.D., Principal Investigator — G.R.M.O. Inc.
Locations (1):
- G.R.M.O. Inc., Québec, Quebec, Canada

REFERENCES:
- [Background] Osteoporosis prevention, diagnosis, and therapy. NIH Consens Statement. 2000 Mar 27-29;17(1):1-45. PMID 11525451
- [Background] Eastell R. Treatment of postmenopausal osteoporosis. N Engl J Med. 1998 Mar 12;338(11):736-46. doi: 10.1056/NEJM199803123381107. No abstract available. PMID 9494151
- [Background] Raisz LG. Clinical practice. Screening for osteoporosis. N Engl J Med. 2005 Jul 14;353(2):164-71. doi: 10.1056/NEJMcp042092. No abstract available. PMID 16014886
- [Background] Dempster DW, Lindsay R. Pathogenesis of osteoporosis. Lancet. 1993 Mar 27;341(8848):797-801. doi: 10.1016/0140-6736(93)90570-7. No abstract available. PMID 8096008
- [Background] Cree MW, Juby AG, Carriere KC. Mortality and morbidity associated with osteoporosis drug treatment following hip fracture. Osteoporos Int. 2003 Sep;14(9):722-7. doi: 10.1007/s00198-003-1430-3. Epub 2003 Aug 7. PMID 12904833
- [Background] Kanis JA, Oden A, Johnell O, De Laet C, Jonsson B, Oglesby AK. The components of excess mortality after hip fracture. Bone. 2003 May;32(5):468-73. doi: 10.1016/s8756-3282(03)00061-9. PMID 12753862
- [Background] Takada Y, Aoe S, Kumegawa M. Whey protein stimulated the proliferation and differentiation of osteoblastic MC3T3-E1 cells. Biochem Biophys Res Commun. 1996 Jun 14;223(2):445-9. doi: 10.1006/bbrc.1996.0913. PMID 8670301
- [Background] Matsuoka Y, Serizawa A, Yoshioka T, Yamamura J, Morita Y, Kawakami H, Toba Y, Takada Y, Kumegawa M. Cystatin C in milk basic protein (MBP) and its inhibitory effect on bone resorption in vitro. Biosci Biotechnol Biochem. 2002 Dec;66(12):2531-6. doi: 10.1271/bbb.66.2531. PMID 12596844
- [Background] Olsson SL, Ek B, Bjork I. The affinity and kinetics of inhibition of cysteine proteinases by intact recombinant bovine cystatin C. Biochim Biophys Acta. 1999 Jun 15;1432(1):73-81. doi: 10.1016/s0167-4838(99)00090-4. PMID 10366730
- [Background] Inaoka T, Bilbe G, Ishibashi O, Tezuka K, Kumegawa M, Kokubo T. Molecular cloning of human cDNA for cathepsin K: novel cysteine proteinase predominantly expressed in bone. Biochem Biophys Res Commun. 1995 Jan 5;206(1):89-96. doi: 10.1006/bbrc.1995.1013. PMID 7818555
- [Background] Yamamura J, Morita Y, Takada Y, Kawakami H. The fragments of bovine high molecular weight kininogen promote osteoblast proliferation in vitro. J Biochem. 2006 Dec;140(6):825-30. doi: 10.1093/jb/mvj217. Epub 2006 Oct 28. PMID 17071946
- [Background] Uenishi K, Ishida H, Toba Y, Aoe S, Itabashi A, Takada Y. Milk basic protein increases bone mineral density and improves bone metabolism in healthy young women. Osteoporos Int. 2007 Mar;18(3):385-90. doi: 10.1007/s00198-006-0228-5. Epub 2006 Oct 18. PMID 17048062
- [Background] Toba Y, Takada Y. [Prevention of osteoporosis by foods and dietary supplements. "Mainichi Hone Kea MBP": A foods for specified health uses (FOSHU) product containing MBP that has an effect to increase bone density]. Clin Calcium. 2006 Oct;16(10):1701-5. Japanese. PMID 17012824
- [Background] Takada Y, Kobayashi N, Kato K, Matsuyama H, Yahiro M, Aoe S. Effects of whey protein on calcium and bone metabolism in ovariectomized rats. J Nutr Sci Vitaminol (Tokyo). 1997 Apr;43(2):199-210. doi: 10.3177/jnsv.43.199. PMID 9219093
- [Background] Toba Y, Takada Y, Yamamura J, Tanaka M, Matsuoka Y, Kawakami H, Itabashi A, Aoe S, Kumegawa M. Milk basic protein: a novel protective function of milk against osteoporosis. Bone. 2000 Sep;27(3):403-8. doi: 10.1016/s8756-3282(00)00332-x. PMID 10962352
- [Background] Kruger CL, Marano KM, Morita Y, Takada Y, Kawakami H, Kobayashi T, Sunaga M, Furukawa M, Kawamura K. Safety evaluation of a milk basic protein fraction. Food Chem Toxicol. 2007 Jul;45(7):1301-7. doi: 10.1016/j.fct.2007.01.017. Epub 2007 Jan 30. PMID 17397980
- [Background] Aoe S, Toba Y, Yamamura J, Kawakami H, Yahiro M, Kumegawa M, Itabashi A, Takada Y. Controlled trial of the effects of milk basic protein (MBP) supplementation on bone metabolism in healthy adult women. Biosci Biotechnol Biochem. 2001 Apr;65(4):913-8. doi: 10.1271/bbb.65.913. PMID 11388472
- [Background] Yamamura J, Aoe S, Toba Y, Motouri M, Kawakami H, Kumegawa M, Itabashi A, Takada Y. Milk basic protein (MBP) increases radial bone mineral density in healthy adult women. Biosci Biotechnol Biochem. 2002 Mar;66(3):702-4. doi: 10.1271/bbb.66.702. PMID 12005077
- [Background] Aoe S, Koyama T, Toba Y, Itabashi A, Takada Y. A controlled trial of the effect of milk basic protein (MBP) supplementation on bone metabolism in healthy menopausal women. Osteoporos Int. 2005 Dec;16(12):2123-8. doi: 10.1007/s00198-005-2012-3. Epub 2005 Aug 31. PMID 16133638
- [Background] Toba Y, Takada Y, Matsuoka Y, Morita Y, Motouri M, Hirai T, Suguri T, Aoe S, Kawakami H, Kumegawa M, Takeuchi A, Itabashi A. Milk basic protein promotes bone formation and suppresses bone resorption in healthy adult men. Biosci Biotechnol Biochem. 2001 Jun;65(6):1353-7. doi: 10.1271/bbb.65.1353. PMID 11471735
- [Background] Shatenstein B, Nadon S, Godin C, Ferland G. Development and validation of a food frequency questionnaire. Can J Diet Pract Res. 2005 Summer;66(2):67-75. doi: 10.3148/66.2.2005.67. PMID 15975195
- [Background] Shatenstein B, et al. Plausability assessment and quality assurance of Food Frequency Questionnaires completed in studies of diet and health International Conference on Diet and Activity Methods (ICDAM) p. 281-282, 2009.
- [Background] Eating well with Canada's Food Guide (c) 2007
- [Background] Canadian Nutrient File. H.W.C. Bureau of Nutriional Sciences, Editor. 1982.
- [Background] Shatenstein B, et al. (and members of the the Division on Nutrition and Healthy Aging, FRSQ Network on Aging), Dietary intakes of homedwelling elderly Quebecers obtained from a food frequency questionnaire: A pilot study. J Nutre Health & Aging 7(4): 234-235, 2003.
- [Background] Yamamura J, Takada Y, Goto M, Kumegawa M, Aoe S. Bovine milk kininogen fragment 1.2 promotes the proliferation of osteoblastic MC3T3-E1 cells. Biochem Biophys Res Commun. 2000 Mar 16;269(2):628-32. doi: 10.1006/bbrc.2000.2326. PMID 10708605
- [Background] Hiddink, J., R. de Bore, and D. Romijin Neth Milk Dairy J 32: p. 80-93, 1978.
- [Background] Takada, Y., et al., Whey protein suppresses the osteoclast-mediated bone resorption and osteoclast cell formation. Int Dairy J 7: 821-825, 1997
- [Background] Takada, Y., et al., Milk whey protein enhances the bone breaking force in ovariectomized rats. Nutr Res 17: 1709-1720, 1997.
- [Background] Kato, K., et al., Milk basic protein enhances the bone strength in ovariectomized rats. J Food Biochem 24:467-478, 2000.
- [Background] Corder, G.W.F., D.I. Nonparametric Statistics for Non-Statisticians: A Step-by-Step Approach. New Jesrsey. Wiley. 2009.